CLINICAL TRIAL: NCT02394665
Title: Phase II Study of Dose Escalated, Targeted Radiation Therapy Using 3D Magnetic Resonance Spectroscopy Imaging (MRSI) in Newly Diagnosed Glioblastoma
Brief Title: Dose Escalated MRSI Guided Radiation Therapy in Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Accrual/Enrollment
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140540
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-11

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Gliosarcoma; GBM
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Intensity-Modulated; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1: SIB + IMRT (Experimental): * Simultaneous Integrated Boost (SIB) plus Fractionated Intensity Modulated Radiation therapy (IMRT), with concurrent Temozolomide therapy for 6 weeks;
  * 3D MRSI during week 3, end of RT and other protocol-defined time points during adjuvant Temozolomide therapy;
  * Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire administered at protocol-defined time points;
  * Adjuvant Temozolomide Therapy for up to 12 cycles.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Temozolomide; Behavioral: Functional Assessment of Cancer Therapy-Brain (FACT-Br); Radiation: Simultaneous Integrated Boost; Device: 3D MRSI
- Group 2: SRS Boost + IMRT (Experimental): For patients with High-Risk Tumor Volumes (HTV) <= 4cm; or multiple HTVs <= 3 cm:
  * Stereotactic Radiosurgery Boost (SRS Boost) followed one week later by Fractionated Intensity Modulated Radiation therapy (IMRT), and concurrent Temozolomide therapy for 6 weeks;
  * 3D MRSI during week 3, end of RT and other protocol-defined time points during adjuvant Temozolomide therapy;
  * Functional Assessment of Cancer Therapy-Brain (FACT-Br) questionnaire administered at protocol-defined time points;
  * Adjuvant Temozolomide Therapy for up to 12 cycles.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Temozolomide; Behavioral: Functional Assessment of Cancer Therapy-Brain (FACT-Br); Radiation: Stereotactic Radiosurgery Boost; Device: 3D MRSI

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — IMRT treatment will consist of 60 Gy in 30 fractions to PTV 60
  Other Names: IMRT; Fractionated RT
Drug: Temozolomide — Concurrently during radiation therapy. Adjuvant therapy administered daily on days 1 - 5 for 12 cycles. One cycle = 28 days:
  * Concurrent during Radiation Therapy: 75 mg/m^2 orally for 6 weeks;
  * Post-radiation, adjuvant therapy: 150 mg/m^2 - 200 mg/m^2 orally daily on days 1 - 5 of each cycle.
  Other Names: Temodar; Temodal
Behavioral: Functional Assessment of Cancer Therapy-Brain (FACT-Br) — FACT-Br Quality of Life (QOL) questionnaire to be completed by study patients as protocol specific timepoints
  Other Names: FACT-Br
Radiation: Stereotactic Radiosurgery Boost — Patients will undergo SRS boost in a single fraction dose prior to IMRT treatment:
  HTV Maximum dimension vs. Prescribed Dose to HTV: ≤ 20 mm = 21 Gy; 21 mm - 30 mm = 18 Gy; 31 mm - 40 mm = 15 Gy.
  Other Names: SRS Boost
  Arms: Group 2: SRS Boost + IMRT
Radiation: Simultaneous Integrated Boost — Treatment shall consist of 60 Gy in 30 fractions to planning target volume (PTV) 60 and 75 Gy in 30 fractions to PTV 75.
  Other Names: SIB
  Arms: Group 1: SIB + IMRT
Device: 3D MRSI — Three Dimensional Magnetic Resonance Spectroscopy Imaging (MRSI) during pre-treatment, week 3 during radiation therapy, end of radiation therapy; will include standard gadolinium enhanced MRI prior to cycle 1, 5, 9, and post cycle 12 of adjuvant temozolomide therapy, per protocol.
  Other Names: 3D Magnetic Resonance Spectroscopy Imaging

SUMMARY:
In summary, the overall prognosis of glioblastoma (GBM) patients remains poor. Although clinical gains have been achieved in the past, these have been modest, with a majority of patients succumbing to local disease progression within 2 years. New strategies for treatment need to be identified which enhance local control above the current treatment regimen in order to achieve further clinical gains in this disease. Favorable early experience with magnetic resonance spectroscopy imaging (MRSI) demonstrates that metabolic imaging can identify active tumor beyond standard MRI as well as high risk regions at risk for local failure. There is also clinical evidence that limited field dose escalation with either simultaneous integrated boost (SIB) or stereotactic radiosurgery (SRS) is feasible and safe. Coupling these findings provide the rationale for this proposed Phase II trial designed to define efficacy and toxicity of the novel treatment approach of whole brain volumetric 3D MRSI guided dose-escalated radiation therapy (RT) in newly diagnosed GBM patients.

DETAILED DESCRIPTION:
This phase II study will investigate efficacy and safety of volumetric 3D MRSI-directed treatment for newly diagnosed GBM patients. This study will enroll 48 patients in order to obtain at least 40 patients receiving RT and temozolomide. Depending on the size and number of HTVs, a patient will receive either simultaneous integrated boost (SIB) with IMRT (Group 1) or SRS boost followed by IMRT 1 week later (Group 2). Duration of enrollment will be 2 years and minimum follow-up will be 2 years.

The duration of treatment and follow-up will occur as follows:

* Six weeks of RT with concurrent Temozolomide treatment;
* 3D MRSI at week 3 and at the end of RT;
* 28 day break;
* Adjuvant treatment with Temozolomide administered daily on days 1-5 of each cycle, for up to 12 cycles (one cycle = 28 days) which will include standard gadolinium enhanced MRI and 3D MRSI prior to cycle 1, 5, 9, and post cycle 12 of adjuvant Temozolomide;
* Active follow-up at least every three months for one year after the end of adjuvant Temozolomide treatment;
* After one year follow-up for survival will occur every three months for one year.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of glioblastoma (WHO grade IV). Since gliosarcoma is a variant of glioblastoma, gliosarcoma is also an eligible diagnosis.
2. The tumor must have a supratentorial component
3. Patients must have recovered from the effects of surgery, postoperative infection and other complications
4. Karnofsky performance status > 70
5. Age > 18 years
6. Adequate bone marrow function defined as follows:

   * Absolute neutrophil count (ANC) >/= 1500 cells/mm^3
   * Platelet count > 100,000 cells/mm^3
   * Hemoglobin > 10.0 g/dL (Note: the use of transfusion or other intervention to achieve Hgb > 10.0 g/dL is acceptable.)
7. Patients on full-dose anticoagulants (e.g., warfarin or low-molecular weight (LMW) heparin) must meet both of the following criteria:

   * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
   * In-range international normalized ratio (INR) (usually between 2 and 3) on a stable dose of oral anticoagulant or on a stable dose of low molecular weight heparin
8. Adequate renal function, defined as follows:

   * Blood urea nitrogen (BUN) < 30 mg/dL
   * Serum creatinine < 1.5 x upper limit of normal (ULN)
9. Adequate hepatic function, as defined below:

   * Bilirubin < 1.5 normal range
   * Alanine transaminase (ALT) < 3x normal range
   * Aspartate transaminase (AST) < 3x normal range
10. Patients must not be pregnant (positive pregnancy test) or breast feeding; pregnancy test must be done within 7 days prior to registration. Effective contraception (men and women) must be used in patients of child-bearing potential while on study treatment and for 6 months after.
11. Ability to understand and the willingness to sign a written informed consent document
12. Ability to have MRI Scans
13. Ability to swallow capsules

Exclusion Criteria:

1. Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity or cervix are all permissible)
2. Recurrent malignant glioma or evidence of leptomeningeal spread
3. Metastases detected below the tentorium or beyond the cranial vault
4. Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment
5. Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation therapy fields
6. Prior radiation therapy or chemotherapy for glioblastoma
7. Severe, active co-morbidity, defined as follows:

   * Symptomatic congestive heart failure of New York heart Association Class III or IV
   * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within the last 6 months, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
   * Severely impaired lung function as defined as spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
   * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
   * Active (acute or chronic) or uncontrolled severe infections requiring intravenous antibiotics
   * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
   * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition or known HIV seropositivity. Note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with HIV/AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
   * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity
   * Other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy
8. Pregnancy
9. Women who are breast feeding
10. Prior allergic reaction to temozolomide
11. Treatment on any other therapeutic clinical protocol
12. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter their absorption of temozolomide (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
13. Contraindications to MRI including but not limited to, pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steelworker or other implants
14. Need to continue treatment with any prohibited medication (e.g. antioxidants) or have not completed the appropriate washout period.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fazilat Ishkanian, MD, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data were not analyzed due to insufficient number of evaluable subjects. Only one subject enrolled who was later withdrawn by the Investigator prior to assignment to any treatment group or receiving any protocol therapy.
Groups:
- No Treatment Group Assigned: For subject withdrawn from study prior to assignment of treatment group. No protocol therapy received.
Period: Overall Study
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT
Started | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data were not analyzed due to insufficient number of evaluable subjects. Only one subject enrolled who was later withdrawn by the Investigator prior to assignment to any treatment group or receiving any protocol therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 1 | 0 | 0 | 1
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Overall Survival (OS) in Study Patients
Description: The efficacy of 3D MRSI-guided, dose escalated radiation in newly diagnosed glioblastoma (GBM) patients as measured by overall survival (OS). Overall survival (OS) is defined as the time elapsed from the start of study treatment until death. Surviving patients (including patients lost to follow up) will be censored at the date of last contact.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Rate of Progression-Free Survival (PFS) in Study Patients
Description: Rate of progression-free survival in study participants. Progression-free survival (PFS) is defined as the time elapsed from the start of study treatment to the date of documented progression events. For progression-free patients (without progression events), PFS will be censored at the last date of documented PF status.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Rate of Grade 3 or Higher Toxicity as a a Consequence of Study Therapy.
Description: Rate of Grade 3 of Higher Toxicity in study participants as a consequence of study therapy.
Time Frame: 2 years
Population: as for baseline characteristics
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Quality of Life From Baseline in Study Participants
Description: Change in quality of life during radiation and across the longitudinal progression-free interval compared to baseline. Change of quality of life will be assessed and scored via the FACT-Br behavioral questionnaire.
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Patterns of Failure in Study Participants Post-Protocol Therapy
Description: Patterns of Failure will be assessed by determining the number of failures that arise in-field compared to the number that arise out-of-field. In-field failure will be defined as those where greater than 80% of the recurrence volume was encompassed by the 95% prescription isodose line. In addition, we will also describe failures by three types: unifocal, multifocal and diffuse (multicentric including leptomeningeal dissemination).
Time Frame: Up to 2 years
Population: as for baseline characteristics
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Data were not analyzed due to insufficient number of evaluable subjects. Only one subject enrolled who was later withdrawn by the Investigator prior to assignment to any treatment group or receiving any protocol therapy.
Arm/Group | No Treatment Group Assigned | Group 1: SIB + IMRT | Group 2: SRS Boost + IMRT
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data were not analyzed due to insufficient number of evaluable subjects. Only one subject enrolled who was later withdrawn by the Investigator prior to assignment to any treatment group or receiving any protocol therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes